CLINICAL TRIAL: NCT05690516
Title: The Protective Effect of Mask Wearing Against Respiratory Tract Infections: a Pragmatic Randomized Trial
Brief Title: The Protective Effect of Mask Wearing Against Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 536544
Record Dates: First submitted 2023-01-11; First posted 2023-01-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Respiratory Tract Infections
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Sequence generation. We will use a simple 1:1 randomization by means of computer-generated random numbers.
  The allocation will be concealed as the participant themselves will be directly informed of their allocation as soon as they have agreed to take part in the trial and have completed the online consent and baseline form. Generation of allocation sequence, enrolment of participants and assignment of participants will all be handled by the digital recruitment platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face masks (Experimental): Participants in the experimental arm are asked to wear face masks when close to others outside their home, e.g., in public spaces like shopping centres, and streets and on public transport.
  Interventions: Behavioral: Wearing face masks
- Not face masks (No Intervention): Participants in the no intervention arm arm are asked not to wear face masks when close to others outside their home, e.g., in public spaces like shopping centres, and streets and on public transport.

INTERVENTIONS:
Behavioral: Wearing face masks — Participants are asked to wear face masks in public spaces.
  Arms: Face masks

SUMMARY:
In this trial the researchers plan to recruit 4,000 volunteers to be randomly allocated either wearing face masks in public spaces where they are close to other people, or not wear face masks in such circumstances. For each participant the trial period is 2 weeks, after which they will be asked to complete a brief questionnaire which includes questions about whether they experienced the common cold, influenzas or COVID-19 symptoms during the trail period.

DETAILED DESCRIPTION:
This study is a pragmatic, two-armed cluster randomized superiority trial including participants in Norway. Participants will be randomized to one of the following two arms: control group or medical masks in a 1:1 ratio. The primary outcome is self-reported respiratory infection.

The intervention is to ask participants in the intervention groups to wear face masks when close to others outside their home, e.g., in public spaces like shopping centres, and streets and on public transport. The control group will be asked not to wear face masks when close to others outside their home, e.g., in public spaces like shopping centres, and streets and on public transport. Participants will continue to use, or not use, face masks at work independent of which group they are allocated to.

The trial will be fully remote and without any personal interaction between investigators and participants.

The researchers aim to include about 4,000 participants to have a statistical power of 80% to detect a relative risk reduction of 30% for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* Are willing to be randomized to wear, or not to wear, face masks outside their home when close to others for a 14-day period
* Provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4575 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Respiratory symptoms of the common cold, influenza or COVID-19 | Day 1 to 17
  Self-report

SECONDARY OUTCOMES:
Covid-19 prevalence | Day 1 to 17
  Self-report
Positive test for SARS-CoV-2 | Day 3 to 17 after start of tiral period
  We will compare the incidence of notified cases of COVID-19 (i.e. registered positive SARS-CoV-tests)
Health care use for respiratory symptoms | Day 1 to 17
  Self-report
Health care use for injuries | Day 1 to 17
  Self-report
Health care use (all causes) | Day 1 to 17
  Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Runar Solberg, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The researchers intend to give full access to the protocol, participant level-data dataset and statistical code to anyone who is interested, after securing that the dataset is fully anonymized.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The investigators expect to be able to share unidentifiable dataset with partners inside the European Union (EU) by May 2023, and an anonymous dataset for wide distribution at a later stage.

REFERENCES:
- [Derived] Solberg RB, Fretheim A, Elgersma IH, Fagernes M, Iversen BG, Hemkens LG, Rose CJ, Elstrom P. Personal protective effect of wearing surgical face masks in public spaces on self-reported respiratory symptoms in adults: pragmatic randomised superiority trial. BMJ. 2024 Jul 24;386:e078918. doi: 10.1136/bmj-2023-078918. PMID 39048132